CLINICAL TRIAL: NCT03938454
Title: A Prospective Phase II, Open-Label, Single-arm, Multicenter, Study to Assess Efficacy and Safety of SEG101 (Crizanlizumab), in Sickle Cell Disease Patients With Priapism (SPARTAN)
Brief Title: A Study to Evaluate the Safety and Efficacy of Crizanlizumab in Sickle Cell Disease Related Priapism
Acronym: SPARTAN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSEG101AUS05
Record Dates: First submitted 2019-05-02; First posted 2019-05-06 (Actual); Results first posted 2025-03-10 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Priapism
Keywords: Priapism; sickle cell disease; SCD; crizanlizumab; P-selectin; SEG101; monoclonal antibody; prolonged erection; painful erection
MeSH Terms: conditions — Priapism; Anemia, Sickle Cell | interventions — crizanlizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Crizanlizumab 5 mg/kg (Experimental): Participants received 5 mg/kg by IV infusion on Week 1 Day 1, Week 3 Day 1, and on Day 1 of every 4-week cycle until Week 51.
  Interventions: Drug: Crizanlizumab

INTERVENTIONS:
Drug: Crizanlizumab — Crizanlizumab is a concentrate for solution for infusion, IV use. Supplied in single use 10 mL vials at a concentration of 10 mg/mL. One vial contains 100 mg of crizanlizumab.
  Other Names: SEG101

SUMMARY:
The goal of the study was to evaluate the efficacy and safety of crizanlizumab in sickle cell disease (SCD) patients with priapism.

DETAILED DESCRIPTION:
Before participating in this study, information to determine key eligibility criteria was collected as a part of a 14-week Pre-Screening period. The study included a 12-week Screening period and a 52-week (1 year) Treatment period. Eligible participants received crizanlizumab 5 mg/kg by intravenous infusion (IV). Study treatment was received at clinic visits on Week 1 Day 1, Week 3 Day 1, and then on Day 1 of every 4-week cycle. Efficacy assessments included evaluation of priapic and vaso-occlusive (VOC) events. Safety assessments included laboratory tests, electrocardiograms (ECGs), vital signs and physical examinations. Participants had a safety follow-up for up to 15 weeks after the last dose.

ELIGIBILITY:
Inclusion criteria

* Male patients aged 12 years and above
* Confirmed diagnosis of SCD by hemoglobin electrophoresis or high-performance liquid chromatography. All SCD genotypes were eligible (HbSS, HbSβ0, HbSC, HbSβ+, and others)
* Experienced 4 or more priapic events (unwanted erection lasting at least 60 minutes) over the 14 weeks preceding study participation
* Experienced at least 3 priapic events (unwanted erection lasting at least 60 minutes) during the 12-week Screening period with at least 1 event occurring within 4 weeks prior to the first treatment
* If receiving hydroxyurea/hydroxycarbamide or L-glutamine or erythropoietin stimulating agent or voxelotor, must have been receiving the drug for at least 14 weeks prior to screening and planned to continue taking the drug at the same dose and schedule during the trial
* If receiving prophylactic treatment for priapism, must have been receiving the drug for at least 14 weeks prior to screening and planned to continue taking the drug at the same dose and schedule during the trial
* Written informed consent (or assent/parental consent for minor participants) prior to any screening procedures

Exclusion criteria:

* Had penile prosthetic implants or shunts or any other surgical procedure on the penis performed within 12 months prior to consenting was not allowed
* Took drugs/medications that may induce priapism over the 14 weeks preceding study entry
* Received leuprolide acetate (Lupron) or any other gonadotropin releasing hormone receptor agonist agent within 3 months before pre-screening
* Had an erection lasting more than 12 hours over the 14 weeks preceding study entry
* Had an erection lasting more than 12 hours during the 12 weeks of the Screening period

Ages: 12 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 36 (Actual)
Dates: Start 2019-10-16 (Actual); Primary Completion 2023-03-28 (Actual); Study Completion 2023-11-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - University Of Alabama, Birmingham, Alabama
  - University of Connecticut Health Center, Farmington, Connecticut
  - Childrens National Hospital, Washington D.C., District of Columbia
  - Foundation for Sickle Cell Disease Research, Hollywood, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - LSU Medical Center, Shreveport, Louisiana
  - Childrens Hosp Boston Dept of Hematology, Boston, Massachusetts
  - Montefiore Medical Center, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - Brody School of Medicine, Greenville, North Carolina
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Prisma Health Upstate, Greenville, South Carolina
  - University of Texas Medical School, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent expert panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2419
- See also: A Pediatric Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/ppatientsummary/ppatientsummaries?periodicPatientSummaryId=677

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Crizanlizumab 5 mg/kg
Started | 36
Completed | 30
Not Completed | 6
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 2
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) included all enrolled participants to whom the study treatment was assigned regardless of whether or not they had received at least one dose of study treatment or had at least one post-baseline assessment.
Arm/Group | Crizanlizumab 5 mg/kg
Number analyzed (Participants) | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.5 (10.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 33
  Unknown or Not Reported | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 36

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Priapic Events From Baseline to 26 Weeks
Description: A priapic event was defined as an unwanted or painful penile erection lasting at least 60 minutes. Priapic events were self-reported via an electronic reporting system, and data was collected throughout the study period. Number of priapic events was summarized at Baseline (adjusted for 26 weeks) and by 26 weeks, and percent reduction from adjusted Baseline by 26 weeks was summarized.
Time Frame: Baseline up to 26 weeks
Population: The full analysis set (FAS) included all enrolled participants to whom the study treatment was assigned regardless of whether or not they received at least one dose of study treatment or had at least one post-baseline assessment.
Measure: Median (Inter-Quartile Range); unit: Percent change from baseline
Arm/Group | Crizanlizumab 5 mg/kg
Number analyzed (Participants) | 36
Percent change from baseline | -61.3 [-80.1 to -17.3]
Statistical Analysis 1: Comparison: Crizanlizumab 5 mg/kg; Test type: Other; p = 0.0676, Wilcoxon Sign Rank Test — P-value is from one-sided Wilcoxon Sign Rank Test with at least 25% percent reduction from Baseline (adjusted for 26 weeks) as outcome variable; Hodges-Lehmann = 45.98, 95% CI 2-sided [23.50 to 65.36]

2. Secondary Outcome: Annualized Rate of Priapic Events
Description: A priapic event was defined as an unwanted or painful penile erection lasting at least 60 minutes. Priapic events were self-reported via an electronic reporting system, and data was collected throughout the study period.
  The annualized rate of events was defined as the total number of events for a participant occurring from the date of initial infusion to the last contact date of the Treatment Phase of the study x 365.25 divided by the number of days during that same time period. The calculation accounted for early dropouts or lost to follow-up by extrapolating the priapism events rate of every participant to 1 year.
Time Frame: Baseline up to 26 and 52 weeks
Population: The FAS included all enrolled participants to whom the study treatment was assigned regardless of whether or not they received at least one dose of study treatment or had at least one post-baseline assessment.
Measure: Median (Inter-Quartile Range); unit: Events per year
Arm/Group | Crizanlizumab 5 mg/kg
Number analyzed (Participants) | 36
Events per year
  Annualized rate of priapic events by 26 weeks | 31.1 [10.2 to 97.4]
  Annualized rate of priapic events by 52 weeks | 25.6 [9.9 to 68.7]

3. Secondary Outcome: Number of Acute Priapic Events From Baseline to 26 and 52 Weeks
Description: An acute priapic event was defined as an unwanted, painful erection that lasted more than 4 hours and required a visit to the emergency room.
Time Frame: Baseline up to 26 and 52 weeks
Population: The FAS included all enrolled participants to whom the study treatment was assigned regardless of whether or not they received at least one dose of study treatment or had at least one post-baseline assessment. Only participants with Acute Priapic Events are included in this analysis.
Measure: Median (Full Range); unit: Number of acute priapic events
Arm/Group | Crizanlizumab 5 mg/kg
Number analyzed (Participants) | 11
Number of acute priapic events
  Number of acute priapic events at Baseline: number analyzed (Participants) | 3
  Number of acute priapic events at Baseline | 7.0 [2 to 11]
  Number of post-baseline acute priapic events by 26 weeks: number analyzed (Participants) | 2
  Number of post-baseline acute priapic events by 26 weeks | 1.5 [1 to 2]
  Number of post-baseline acute priapic events by 52 weeks: number analyzed (Participants) | 8
  Number of post-baseline acute priapic events by 52 weeks | 1.0 [1 to 2]

4. Secondary Outcome: Annualized Rate of Uncomplicated Vaso-occlusive Crises (VOCs)
Description: An uncomplicated VOC event was defined as an acute event of pain with no known cause for pain other than a VOC event; and requiring treatment with a parenteral or oral opioids or other parenteral analgesic; but was NOT classified as an acute chest syndrome, hepatic sequestration, splenic sequestration or priapism. Events included both healthcare and self-reported events.
  The annualized rate of events was defined as the total number of events for a participant occurring from the date of initial infusion to the last contact date of the Treatment Phase of the study x 365.25 divided by the number of days during that same time period. The calculation accounted for early dropouts or lost to follow-up by extrapolating the priapism events rate of every participant to 1 year.
Time Frame: Baseline up to 26 and 52 weeks
Population: The FAS included all enrolled participants to whom the study treatment was assigned regardless of whether or not they received at least one dose of study treatment or had at least one post-baseline assessment. Only participants who had uncomplicated VOC events within the specified time frame were included in the analysis.
Measure: Median (Inter-Quartile Range); unit: Events per year
Arm/Group | Crizanlizumab 5 mg/kg
Number analyzed (Participants) | 24
Events per year
  Annualized rate of uncomplicated VOCs by 26 weeks: number analyzed (Participants) | 18
  Annualized rate of uncomplicated VOCs by 26 weeks | 4.1 [3.9 to 8.0]
  Annualized rate of uncomplicated VOCs by 52 weeks | 2.5 [1.4 to 6.8]

5. Secondary Outcome: Annualized Rate of Complicated VOCs
Description: Complicated VOCs were defined as acute chest syndrome, hepatic sequestration, splenic sequestration, and acute priapism recorded by healthcare visit.
  The annualized rate of events was defined as the total number of events for a participant occurring from the date of initial infusion to the last contact date of the Treatment Phase of the study x 365.25 divided by the number of days during that same time period. The calculation accounted for early dropouts or lost to follow-up by extrapolating the priapism events rate of every participant to 1 year.
Time Frame: Baseline up to 26 and 52 weeks
Population: The FAS included all enrolled participants to whom the study treatment was assigned regardless of whether or not they received at least one dose of study treatment or had at least one post-baseline assessment. Only participants who had complicated VOC events within the specified time frame were included in the analysis.
Measure: Median (Inter-Quartile Range); unit: Events per year
Arm/Group | Crizanlizumab 5 mg/kg
Number analyzed (Participants) | 2
Events per year
  Annualized rate of complicated VOCs by 26 weeks: number analyzed (Participants) | 1
  Annualized rate of complicated VOCs by 26 weeks | 1.9 [1.9 to 1.9]
  Annualized rate of complicated VOCs by 52 weeks | 1.4 [0.9 to 1.9]

6. Post Hoc Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) Associated With Infusion Related Reactions (Adverse Events of Special Interest)
Description: A TEAE was defined as an adverse event starting or worsening after the administration of study medication. TEAEs experienced by participants in association with infusion related reactions were classified as adverse events of special interest (AESIs).
Time Frame: Baseline up to 57 weeks
Population: The Safety Analysis Set consisted of all participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Crizanlizumab 5 mg/kg
Number analyzed (Participants) | 36
Participants
  With at least one AESI | 9
  Axillary pain | 1
  Non-cardiac chest pain | 1
  Infusion related reaction | 2
  Arthralgia | 1
  Back pain | 1
  Neck pain | 1
  Headache | 3
  Pruritis | 1
  Rash maculo-papular | 1

7. Post Hoc Outcome: Percent Change in Priapic Events From Baseline to 26 Weeks Without the Outlier
Description: A priapic event was defined as an unwanted or painful penile erection lasting at least 60 minutes. Priapic events were self-reported via an electronic reporting system, and data was collected throughout the study period. Number of priapic events was summarized at Baseline (adjusted for 26 weeks) and by 26 weeks, and percent reduction from adjusted Baseline by 26 weeks was summarized.
  For one participant, the outlier, a large amount of data corresponding to 38 days of screening (45% of the period), was not reported. Additionally, data in the other days of the Screening Period were also not collected. This was a unique occurrence which did not happen with other participants. To understand its impact, the primary endpoint has also been analyzed excluding this outlier in a post-hoc sensitivity analysis.
Time Frame: Baseline up to 26 weeks
Population: The FAS included all enrolled participants to whom the study treatment was assigned regardless of whether or not they received at least one dose of study treatment or had at least one post-baseline assessment. Analysis was performed excluding one outlier participant, who had a large amount of data unreported.
Measure: Median (Inter-Quartile Range); unit: Percent change from baseline
Arm/Group | Crizanlizumab 5 mg/kg
Number analyzed (Participants) | 35
Percent change from baseline | -63.3 [-81.1 to -17.6]
Statistical Analysis 1: Comparison: Crizanlizumab 5 mg/kg; Test type: Other; p = 0.0259, Wilcoxon Sign Rank Test — P-value is from one-sided Wilcoxon Sign Rank Test with at least 25% reduction from Baseline (adjusted for 26 weeks) as outcome variable; Hodges-Lehmann = 50.20, 95% CI 2-sided [27.94 to 67.36]

ADVERSE EVENTS:
Time Frame: Adverse events were reported from first dose of study treatment until end of study treatment, up to a maximum duration of 57 weeks.
Description: The Safety Analysis Set consisted of all participants who received at least 1 dose of study treatment.
Arm/Group | Crizanlizumab 5 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/36
Serious Adverse Events (participants affected / at risk) | 7/36
Other Adverse Events (participants affected / at risk) | 26/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Crizanlizumab 5 mg/kg (N=36)
Peripheral swelling (General disorders) | 1
Periorbital cellulitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Jugular vein thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Crizanlizumab 5 mg/kg (N=36)
Sinus bradycardia (Cardiac disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 2
Chest discomfort (General disorders) | 2
Fatigue (General disorders) | 3
Non-cardiac chest pain (General disorders) | 2
Pyrexia (General disorders) | 6
COVID-19 (Infections and infestations) | 5
Infusion related reaction (Injury, poisoning and procedural complications) | 2
Amylase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 2
Blood bilirubin increased (Investigations) | 2
Blood creatine phosphokinase increased (Investigations) | 2
Blood lactate dehydrogenase increased (Investigations) | 2
Lymphocyte count increased (Investigations) | 3
Neutrophil count decreased (Investigations) | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 2
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2
Headache (Nervous system disorders) | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 2

LIMITATIONS AND CAVEATS:
This was a single-arm trial in a disease where clinical history has significant variability.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-12-16): https://cdn.clinicaltrials.gov/large-docs/54/NCT03938454/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-20): https://cdn.clinicaltrials.gov/large-docs/54/NCT03938454/SAP_001.pdf